CLINICAL TRIAL: NCT07099183
Title: Nyx3 Eye Mask Physiological Data Collection Study
Brief Title: Nyx3 Data Collection Study
Status: Not yet recruiting | Type: Observational
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Other Study IDs: SLP-25-06-01
Record Dates: First submitted 2025-06-24; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Sleep Staging
Keywords: EEG; Sleep Eye Mask

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nyx3 and Hypnodyne EEG and accelorometer data collection: Participants will use both the Nyx3 eye mask and Hypnodyne headband concurrently in a real-world home sleep environment.

SUMMARY:
Each participant will wear the Nyx3 eye mask and Hypnodyne headband for 1 night at-home. Objectives include collecting and evaluating data quality from the Nyx3 eye mask, and exploring the impact of its paced breathing feature on sleep onset latency.

DETAILED DESCRIPTION:
The Nyx3 data collection study evaluates the Nyx3 EEG eye mask, a wearable device designed to collect EEG data for sleep staging. Traditional sleep diagnostics via polysomnography (PSG) are resource-intensive and limited to clinical settings. This study addresses the need for scalable, home-based, non-invasive sleep monitoring solutions by collecting data for algorithm development and validating the Nyx3 device's feasibility and performance against the Hypnodyne headband-a validated wearable EEG comparator.

60 participants who meet the inclusion criteria will perform the following: Visit 1 Participants will provide written informed consent. Participants will be shown the Nyx3 eye mask and Hypnodyne and shown how to use them and trial them for fit and comfort. If the participant and assessor are happy to proceed, the participants will take the eye mask home to trial.

Visit 2 The participant will return the Nyx3 eye mask to the assessor. The participants' questionnaire responses will be reviewed. This concludes participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants willing to give written informed consent
* Participants who ≥ 18 years of age
* Participants who can trial the eye mask overnight

Exclusion Criteria:

* Participants with active medical implants that interact with magnets (i.e., pacemakers, implantable cardioverter defibrillators (ICD), neurostimulators, cerebrospinal fluid (CSF) shunts, insulin/infusion pumps).
* Participants with metallic implants/objects containing ferromagnetic material (i.e., aneurysm clips/flow disruption devices, embolic coils, stents, valves, electrodes, implants to restore hearing or balance with implanted magnets, ocular implants, metallic splinters in the eye)
* Participants who are or may be pregnant
* Participants who are currently enrolled in other clinical studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be healthy adult volunteers, aged 18 or above, with self-reported normal sleep patterns. The study population will include a diverse sample across age, sex, race, and ethnicity.
  Recruitment strategies will include outreach to both internal and external community participants to ensure a broad representation.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
sleep-related EEG and accelerometry data | Day 1
  The primary endpoint of this study is to evaluate the performance of the Nyx3 eye mask in capturing sleep-related EEG and accelerometry data suitable for automated sleep staging (Night-level summary statistics-such as total sleep time (TST), sleep onset latency (SOL), and percentage time spent in each sleep stage (e.g., %REM, %N3)), and to compare its signal quality and staging outputs against a validated comparator device, the Hypnodyne headband Nyx3. In this study, the primary endpoint is the agreement between the Nyx3 and Hypnodyne sleep-stage labels, which will be captured using Cohen's κ.

SECONDARY OUTCOMES:
Subjective sleep latency | Baseline
  The secondary endpoint of this study is to explore whether the use of the paced breathing feature within the Nyx3 EEG eye mask is associated with subjective reduced sleep onset latency (SOL) and/or improved subjective sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Wimms, PhD, Principal Investigator — ResMed

IPD SHARING:
Plan to Share IPD: No